CLINICAL TRIAL: NCT06798597
Title: Health4Life: A Digital Intervention to Promote Healthy Lifestyle Behaviours From the Start of Life: Protocol for a Hybrid Effectiveness-implementation Study
Brief Title: Health4Life a Digital Intervention to Promote Healthy Lifestyle Behaviours From the Start of Life
Acronym: Health4Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Forte (Industry)
Responsible Party: Principal Investigator, Christine Delisle Nyström, Assistant Professor, Docent, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-07372-01
Record Dates: First submitted 2025-01-20; First posted 2025-01-29 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: Lifestyle behaviours; Childhood

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Health4Life app (Experimental): Receives the Health4Life app for 16 months
  Interventions: Behavioral: Health4Life app
- Usual care (No Intervention): Receives standard care through child healthcare

INTERVENTIONS:
Behavioral: Health4Life app — Health4Life is a program based on the anticipatory guidance approach aiming to support parents create healthy lifestyle behaviours starting in early infancy. The intervention consists of ten themes over a 16 month period and incorporates interactive features such as quizzes.
  Arms: Health4Life app

SUMMARY:
The overall aim of this project is to evaluate the effectiveness and implementation of a digital intervention to support parents to create healthy lifestyle behaviours from the start of their infant's life, in order to prevent overweight and obesity. Using a randomized controlled trial with a hybrid type I implementation-effectiveness design we will:

1. evaluate the effectiveness of the 16-month Health4Life intervention on:

   1. Children's' dietary intake, screen time, physical activity, and sleep
   2. Children's body mass index (BMI) z-scores
   3. Parental self-efficacy
2. Evaluate the cost-effectiveness of the Health4Life app.
3. Evaluate and explore the implementation of the Health4Life app within primary child healthcare with regards to its:

   1. acceptability, appropriateness, and feasibility according to child healthcare nurses.
   2. satisfaction and usage by parents.

ELIGIBILITY:
Inclusion Criteria:

* 0-2 month old infants at routine visits at selected child healthcare centers in Sweden.

Exclusion Criteria:

* Infants diagnosed with a neurological or endocrine disorder.
* Infants who have a parent suffering from a serious physical or psychological disease making the study too demanding for the family.
* Infants from families who will not be able understand the content of the app.

Ages: 0 Months to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 504 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-03-17 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Intake of key dietary indicators | Post-intervention (i.e., 16 months after baseline)
  Intake of dietary indicators such as fruit, vegetables, sweet snacks, savoury snacks, and sugar sweetened beverages (portions or grams per day)
Screen time | Baseline, mid-intervention (i.e., 8 months after baseline), and post-intervention (i.e., 16 months after baseline)
  Time spent watching screens (min/day)
Total physical activity | Post-intervention (i.e., 16 months after baseline)
  Total number of minutes spent in physical activity (min/day) assessed with accelerometers.
Sleep | Post-intervention (i.e., 16 months after baseline)
  Total amount of time spent sleeping (min/day) measured with accelerometers.

SECONDARY OUTCOMES:
BMI | Post-intervention (i.e., 16 months after baseline)
  weight (kg) / height (m)^2
Parental self-efficacy to promote healthy diet and physical activity behaviours in their child | Baseline, mid-intervention (i.e., 8 months after baseline), and post-intervention (i.e., 16 months after baseline)
  Parental self-efficacy for promoting healthy physical activity and dietary behaviours in children scale questionnaire. Minimum score = 0, Maximum score = 160, a better score indicates a better outcome
Satisfaction of the app (Questionnaire) | Post-intervention (i.e., 16 months after baseline)
  Questionnaire to all parents in the intervention group
Satisfaction of the app (Interviews) | Post-intervention (i.e., 16 months after baseline)
  Semi-structured interviews with parents
Usage of the app (Questionnaire) | Post-intervention (i.e., 16 months after baseline)
  Questionnaire to all parents in the intervention group
Usage of the app (Interviews) | Post-intervention (i.e., 16 months after baseline)
  Semi-structured interviews with parents
Accetability of the app | Post-intervention (i.e., 16 months after baseline)
  Semi-structured interviews with child healthcare nurses
Approritateness of the app | Post-intervention (i.e., 16 months after baseline)
  Semi-structured interviews with child healthcare nurses
Feasibility of the app | Post-intervention (i.e., 16 months after baseline)
  Semi-structured interviews with child healthcare nurses
Usage of app by parents (measured objectively through the app) | Post-intervention (i.e., 16 months after baseline)
  Number of times they went in the app, number of read messages, and number of quizzes completed.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Delsile Nyström, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: No